CLINICAL TRIAL: NCT07313163
Title: Evaluation of the Effect of Music During Nursing Care on the Confort of Patient Hospitalized in Intensive Care Unit During the Acute Phase of a Stroke
Acronym: MELODHYA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 778_MELODHYA
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: stroke; nursing care; music
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator)
  Interventions: Other: SOC (Standard of care)
- Music (Experimental)
  Interventions: Other: Use of music during nursing care

INTERVENTIONS:
Other: Use of music during nursing care — during hospitalization for stroke, nursing care will be performed while listening to music
  Arms: Music
Other: SOC (Standard of care) — Nursing care during hospitalization for stroke will be performed as the usual
  Arms: Standard of care

SUMMARY:
Nurses in Stroke Units and Neurovascular Intensive Care Units (USINV) provide care for patients who have experienced a stroke, a sudden and often devastating event that can result in motor, sensory, visual, cognitive, language, or swallowing impairments. Despite advances in stroke management, it remains the leading cause of acquired disability and the second leading cause of death in France, with 122,422 hospitalizations in 2022 and 773 at our institution in 2023. Acute stroke care guidelines recommend hospitalization in specialized neurovascular intensive care units (USINV), as this setting improves survival and recovery through specialized nursing care, close monitoring, and prevention of complications. However, the sudden onset of disability and the unfamiliar, often stressful hospital environment can lead to anxiety, fear, and a sense of helplessness among patients.

Providing comfort is a key nursing objective in this context. Kolcaba defines comfort as the experience of having fundamental needs for relief, well-being, and transcendence met in physical, psycho-spiritual, environmental, and sociocultural dimensions. Hygiene care, in particular, can contribute to comfort by ensuring cleanliness, minimizing pain, and improving self-image. The use of music during care has been proposed as a means to enhance comfort by positively influencing both physical and psychological states, as well as the care environment. Music can stimulate the senses, redirect attention, evoke pleasant memories, reduce stress, and provide a sense of control and identity for patients.

While music therapy-a specialized practice requiring trained professionals-has been studied in various fields, the use of music during routine care is distinct and has shown benefits in psychiatry, palliative care, and geriatrics, as well as during stressful procedures. In stroke rehabilitation, music has been explored for its effects on mood and recovery, but its use during the acute phase of stroke in USINV has not been systematically studied. An informal survey at our institution revealed that 78% of nurses and nursing assistants use music during care, particularly during hygiene procedures.

Our hypothesis is that incorporating music into hygiene care can improve patient comfort by addressing physical, psychological, and environmental needs. To assess comfort in a population that may have communication difficulties, we developed a visual comfort scale (0-5) using artificial intelligence-generated facial expressions. This scale was tested on 30 USINV patients and found to be accessible and easy to use, except for those with cognitive impairments or language barriers, who will be excluded from further study.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking patient
* Aged 18 years or older
* Diagnosed with a stroke
* Hospitalized in a Neurovascular Intensive Care Unit (USINV)
* Requiring a complete bed bath by a nurse or nursing assistant
* Affiliated with a health insurance scheme
* Having provided free, informed, and explicit consent

Exclusion Criteria:

* Patient hospitalized for a reason other than stroke
* Patient with comprehension disorders (aphasia with impaired comprehension, cognitive disorders predating the stroke, confusion, non-French-speaking)
* Blind patient
* Patient under guardianship or curatorship
* Patient deprived of liberty or under legal protection (sauvegarde de justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Auto _ Evaluation of patient confort during nursing care | Day 1
  After the nursing care, Patient will evaluate their confort using a visual confort scale with 5 faces showing extreme discomfort (coded 1) to full confort (coded 5)

SECONDARY OUTCOMES:
Hetero evaluation of patient pain | day 1
  nurses will evaluate patient pain after nursing care using the algoplus scale (0 indicating no pain at all, 30 maximum pain )

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Paris Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No